CLINICAL TRIAL: NCT00298064
Title: Assessment of EGFR Genomic Alterations as Prognostic Markers in Cervical Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0548C
Record Dates: First submitted 2006-02-28; First posted 2006-03-01 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Cervical Cancer; Cervix
Keywords: Cervical cancer; EGFR; cervical; genomic; DNA; markers; prognostic; gene; epidermal growth factor
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Tissue Banks

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Tissue Repository

SUMMARY:
The Tissue Repository will search for cases, pull slides, Paraffin-embedded tissue (PET) blocks.

DETAILED DESCRIPTION:
This study is done to gather preliminary data for determining the best way to test EGFR expression in patients with cervical cancer who will receive treatment with EGFR inhibitors in the future.

This study is designed to obtain preliminary data of genomic and phenotypic alterations of the EGFR pathway in high grade cervical intraepithelial lesions (HG-SIL) and invasive cervical cancers (CC) to be used later for therapeutic guidance and to evaluate genomic (over-expression, amplification, point mutations, etc.) and phenotypic alterations of other transduction pathways interacting with the EGFR pathway.

ELIGIBILITY:
Inclusion Criteria:

* Samples from patients diagnosed with HG-SIL (n=300) and CC (n=300) with a follow-up of at least 24 months, existing at the Department of Pathology will be retrieved by the Tissue Repository, de-identified them and provided with code numbers that will not be linked to patient's data.

Exclusion Criteria:

* None Specified.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-12 (Actual); Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claire Verschraegen, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States